CLINICAL TRIAL: NCT00561834
Title: Ranibizumab Therapy for Non-arteritic Ischemic Optic Neuropathy (NAION)
Brief Title: Ranibizumab Therapy for Non-arteritic Ischemic Optic Neuropathy
Acronym: NAION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0446; genentech FVF4256s (Other: genentech)
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-08

CONDITIONS: Nonarteritic Anterior Ischemic Optic Neuropathy
Keywords: non-arteritic ischemic optic neuropathy; ranibizumab; naion
MeSH Terms: conditions — Optic Neuropathy, Ischemic | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Experimental): To determine the mean change in best corrected visual acuity (BCVA) using the Early Treatment Diabetic Retinopathy Study testing system at 6 months in NAION patients treated as needed (PRN) with ranibizumab.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — All patients (n=15) will be treated with open label 0.5mg ranibizumab given intravitreally monthly as needed for 6 months.

SUMMARY:
The purpose of this study is to explore the safety and efficacy of ranibizumab to treat non-arteritic ischemic optic neuropathy based on clinical and anatomical findings.

DETAILED DESCRIPTION:
Nonarteritic anterior ischemic optic neuropathy (NAION) is the most common acute optic neuropathy in people older than 50 years. It is characterized by sudden partial loss of vision in one eye and has an increased risk of vision loss in the fellow eye. Although cause has not been determined, NAION is thought to occur following an idiopathic ischemic event involving the short posterior ciliary arteries that supply blood to the most anterior part of the optic nerve. A complete loss of vision is rare, but partial loss of visual field or acuity can result from NAION in the affected eye(s).

Patients who have a 'disc at risk' or 'crowded disc' (small cup: disc ratio) are at increased risk for developing NAION. Other risk factors for NAION include age > 50 years and white race (estimated 95% of cases). Hypertension and diabetes also predispose to NAION development. Other factors that have been associated with NAION include high cholesterol, arteriosclerosis, stroke, cardiac and intraocular surgery, tobacco use, nocturnal hypotension, blood loss, glaucoma, elevated homocysteine and sleep apnea. The association between NAION and hypertension, high cholesterol and diabetes is stronger in individuals younger than 50 years than in older persons.

Patients with NAION caused by ischemia leading to swelling of the optic nerve and rapidly progressing visual loss have had limited results with therapy such as corticosteroids, brimonidine, levodopa or surgery, such as optic nerve sheath decompression, in the past. Currently, there is no standard of care for these patients.

Although the role of vascular endothelial growth factor (VEGF) in NAION has not been established, ischemic conditions may lead to VEGF production which could be the cause of edema and swelling. This possibility suggests that VEGF may be a target for therapeutic intervention by ranibizumab. Ranibizumab has demonstrated an effect on edema and vascular permeability. In animal studies it has shown a concentration- dependent effect of blunting the vascular permeability induced by VEGF. Of the more than 5,000 subjects with age-related macular degeneration in current and completed clinical trials, vascular permeability and edema have decreased with the use of ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent
* 21 years of age or older
* new onset, within 14 days, of ischemia and vision loss
* Best Corrected Visual Acuity (BCVA) 20/40 or worse

Exclusion Criteria:

* pregnancy or lactation
* proliferative diabetic retinopathy,
* diabetic macular edema,
* uveitis,
* history of ocular trauma,
* severe glaucoma,
* age-related macular degeneration.
* prior or concomitant treatment of oral steroids within 30 days,
* participation in any studies of investigational drugs within 30 days,
* participation in a ranibizumab clinical trial or,
* prior treatment intravitreally or intravenously of Avastin or steroids.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Mandava, MD, Principal Investigator — Rocky Mountain Lions Eye Institute, University of Colorado Health Sciences Center
Locations (1):
- Rocky Mountain Lions Eye Institute, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: ranibizumab: 0.5mg ranibizumab given intravitreally as needed after initial treatment
Period: Overall Study
Arm/Group | Ranibizumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (4.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity
Description: The mean change in best corrected Snellen visual acuity at 6 months in NAION patients treated as needed with ranibizumab.
Time Frame: Baseline and 6 months
Measure: Number; unit: lines change in Snellen chart
Arm/Group | Ranibizumab
Number analyzed (Participants) | 2
lines change in Snellen chart
  lines change in visual acuity subject 1 | 4
  lines change in visual acuity -subject 2 | 3

ADVERSE EVENTS:
Time Frame: 1 year 5 months
Arm/Group | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes